CLINICAL TRIAL: NCT03891667
Title: Disulfiram ("Antabuse"): A Test of Symptom Reduction Among Patients With Previously Treated Lyme Disease
Brief Title: Disulfiram: A Test of Symptom Reduction Among Patients With Previously Treated Lyme Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Collaborators: FDC Foundation (Other)
Responsible Party: Principal Investigator, Brian A Fallon, Professor of Clinical Psychiatry, Research Foundation for Mental Hygiene, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7755
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Results first posted 2023-06-05 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Fatigue; Quality of Life
Keywords: Lyme Disease; Post-treatment Lyme Disease Syndrome; Disulfiram; Chronic Lyme Disease
MeSH Terms: conditions — Fatigue; Lyme Disease; Post-Lyme Disease Syndrome | interventions — Disulfiram

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to one of two groups:
  Treatment Group I- patients will receive Disulfiram for 8 weeks
  Treatment Group 2 - patients will receive Disulfiram for 4 weeks followed by 4 weeks of placebo.
  The dosing follows a fixed-flexible schedule. Clinical judgment guides dosing increases, based on patient tolerance, side effects, and response.
  Week 1: 250 mg every other day. Week 2: 250 mg daily (or continuation of lower dose based on clinical judgment).
  Week 3: 250 mg alternating with 500 mg/daily (or continued lower dose based on clinical judgment) Week 4: 500 mg daily (or continued lower dose based on clinical judgment)
  Week 5-8: 500 mg/daily (or continued lower dose based on clinical judgment) :
  Primary outcome is at week 10. Patients will be reassessed at week 14.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a placebo-controlled study using matching capsules for disulfiram and placebo. Neither the participant, the care provider, nor the investigator will know the randomized assignment. The research pharmacy and a researcher not involved with this study will keep the code regarding group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 8 Week Disulfiram (Experimental): Patients in this group receive disulfiram for 8 weeks. The dosing schedule is fixed-flexible, starting at 250 mg every other day at week 1, 250 mg daily for week 2, 250 mg alternating with 500 mg for week 3, and 500 mg daily for week 4 to week 8. Dose increases are based on clinical judgment guided by patient tolerance, response, body weight, and side effects.
  Interventions: Drug: Disulfiram
- 4 Week Disulfiram (Active Comparator): Patients in this group receive disulfiram for 4 weeks followed by placebo capsules for 4 weeks. The dosing schedule is fixed-flexible, starting at 250 mg every other day at week 1, 250 mg daily for week 2, 250 mg alternating with 500 mg during week 3, and 500 mg daily during week 4. Placebo capsules are given during weeks 5-8. Dose increases are based on clinical judgment guided by patient tolerance, response, body weight, and side effects.
  Interventions: Drug: Disulfiram

INTERVENTIONS:
Drug: Disulfiram — Patients will receive disulfiram for 4 weeks followed by placebo for 4 weeks or disulfiram for 8 weeks.
  Other Names: Antabuse

SUMMARY:
Approximately 10-20% of patients experience ongoing symptoms despite having received standard antibiotic therapy for Lyme disease. Possible explanations for persistent symptoms include persistent infection and/or post-infectious causes. Recent in vitro studies indicate that disulfiram is effective at killing both the actively replicating and the more quiescent persister forms of Borrelia burgdorferi, the microbe that causes Lyme Disease. In this study, the investigators are examining the safety of disulfiram among patients with post-treatment Lyme disease symptoms. The investigators are also conducting a preliminary investigation regarding the relative benefit of 4 vs 8 weeks of treatment with disulfiram.

DETAILED DESCRIPTION:
Lyme disease, caused by the spirochete Borrelia burgdorferi, is the most common tick-borne illness in the United States. Typically, after being bitten by an infected tick, patients will notice an expanding rash and flu-like symptoms. Most patients recover fully after initial treatment with antibiotics such as doxycycline or amoxicillin. Some patients, however, do not recover fully or their symptoms return within a few months after having completed antibiotic treatment. Common persistent symptoms include fatigue, joint pain, muscle pain, numbness, tingling, burning pains, and changes in mood, memory or mental clarity. These symptoms can last months to years after treatment and, when accompanied by functional impairment, are collectively referred to by the academic community as "Post Treatment Lyme Disease Syndrome (PTLDS)". Patients however typically refer to this constellation of persistent symptoms as "Chronic Lyme Disease".

There are several possible explanations for why patients may have persistent symptoms, including persistent infection and post-infectious changes triggered by the prior infection.

Scientists recently discovered that disulfiram is effective in the lab setting at killing the microbes that cause Lyme disease. Disulfiram is more commonly known as "Antabuse". It is an FDA-approved compound used to assist alcoholics in resisting alcohol consumption. Most remarkable is that disulfiram was effective at killing not only the actively replicating Lyme bacteria (ie, the ones that are typically killed by several antibiotics) but also the relatively dormant or quiescent Lyme bacteria (these are called "drug-tolerant persisters") - these latter spirochetes are the ones that may account for the development of chronic Lyme disease symptoms.

This initial pilot study will focus on patients with persistent symptoms despite having received the standard antibiotic therapy (or more) for Lyme disease. Because no one has yet studied the safety of disulfiram for patients with a history of Lyme disease and because the investigators do not know the optimal treatment duration for disulfiram, the initial effort will have the primary aims of assessing safety and determining whether a longer course of daily treatment is more effective than a shorter course of daily treatment.

The investigators propose therefore a small 14-week randomized placebo-controlled pilot study enrolling 24 patients with persistent symptoms despite prior antibiotic treatment for Lyme disease (known as Post-treatment Lyme Disease Syndrome). Among the 24 disulfiram-treated patients, half will get 8 weeks of disulfiram and the other half will get a shorter duration of disulfiram for 4 weeks followed by 4 weeks of matching placebo. After week 8, patients will be off pills for 2 weeks for the primary week 10 evaluation and then for another 4 weeks for the week 14 follow-up evaluation. This will be a double-blinded study; neither physician nor patient will know which treatment group the patient is assigned to.

With this initial study, the investigators will be able to evaluate the side effects, tolerability and initial signs of the effectiveness of disulfiram in reducing symptoms among the 24 patients assessed. The results of this study will guide the investigators regarding whether a larger definitive randomized trial should be conducted and which treatment schedule is optimal.

ELIGIBILITY:
Inclusion Criteria:

* History of Lyme Disease diagnosis within the prior 16 years History of prior diagnosis of Lyme disease that met the Centers for Disease Control (CDC) surveillance criteria case definition

  * For erythema migrans (EM) rash, this has to be health-care provider diagnosed;
  * For later stages of Lyme disease, this requires a diagnosis of LD by a health-care provider and laboratory testing that confirms a positive result historically.
* History of treatment for Lyme disease that consists of at least 5 weeks of antibiotics (total adding all treatment courses) within the last 16 years.
* Partial Prior Response. History of at least partial response to prior antibiotic therapy for Lyme disease.
* Antibiotic-free interval. Willingness to be off of other antibiotics during the course of this study and for at least 3 months prior to study randomization and during the 14 weeks of this study.
* Current moderate to severe fatigue. The following criteria need to be met:

  1. at least moderate intensity at study screening and at intake (a score of 4 or more on the Fatigue Severity Scale)
  2. triggered or perpetuated by Lyme disease and persisting for at least 6 months after treatment
  3. is not better attributed to another independent medical or psychiatric condition
  4. current episode of Lyme disease-related fatigue is relatively persistent and has not had an intervening interval of 8 months without fatigue since diagnosis of Lyme disease.
* Current post-Lyme symptoms impair the patient's quality of life
* Keeping other current treatments stable- Patients can stay on other non-antibiotic medications as long as these medications have been stable for the 3 months prior to study onset and the dosage regimen does not change during the course of this study (unless the latter is medically or psychiatrically indicated).
* Between the ages 18-65
* Ability to read and speak English

Exclusion Criteria:

* History of cardiovascular disease (e.g., coronary artery disease or heart failure).
* History of seizure disorder, abnormal EEGs, traumatic brain injury, renal disease (e.g. nephritis), liver disease (e.g., hepatitis, CIRRHOSIS), diabetes mellitus, hypothyroidism and/or psychosis. Patients with a history of large fiber neuropathy (EMG/NCS documented) will also be excluded.
* History of Substance Use Disorder (e.g., alcohol abuse, multi-drug dependence) within the past 2 years
* History in the last 6 months of heavy alcohol use which is defined as binge drinking more than 5 days in a one-month period. A binge-drinking episode refers to the consumption of 5 or more drinks for men or 4 or more drinks for women in a 2-hour period.
* Evidence of current active tick-borne illness other than Lyme disease. (Note: patients with evidence of positive antibodies for another TBI will be eligible unless there is evidence that this other TBI is currently active (eg., elevated LFTS (AST & ALT not greater than 2 times upper limit), low platelets, low WBC, high fevers)
* Unwillingness to confirm that he/she will abstain from alcohol and products that may contain alcohol (including sauces, cough syrup, vinegar, backrub products, aftershave lotions) during the month prior to randomization, during the course of this study, and for 6 weeks after the last dose of study medication.
* Inability to confirm abstinence from cannabis or CBD or THC-containing products
* Women who are breastfeeding, pregnant, or at risk of becoming pregnant during the course of the study.
* Patients who are taking or plan to take warfarin, metronidazole, paraldehyde, phenytoin, theophylline, oral anticoagulants, or isoniazid
* A concurrent or recent illness that may better account for current fatigue
* Unwillingness to not take any new non-emergency medications during the course of this study without first reviewing with the study research physician
* History of rubber-contact dermatitis or allergy to disulfiram or thiuram derivatives
* Prior history of serious adverse reaction to disulfiram
* Cognitive Impairment for patients over 60.
* Suicidal acts in the last 6 months or current suicidal thoughts with intent or plan or history of bipolar disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2021-11-26 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian A Fallon, MD, Principal Investigator — Columbia University
Locations (1):
- Lyme Research Center New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There no current plan for sharing participant data.

REFERENCES:
- [Background] Long TE. Repurposing Thiram and Disulfiram as Antibacterial Agents for Multidrug-Resistant Staphylococcus aureus Infections. Antimicrob Agents Chemother. 2017 Aug 24;61(9):e00898-17. doi: 10.1128/AAC.00898-17. Print 2017 Sep. PMID 28674046
- [Background] Pothineni VR, Wagh D, Babar MM, Inayathullah M, Solow-Cordero D, Kim KM, Samineni AV, Parekh MB, Tayebi L, Rajadas J. Identification of new drug candidates against Borrelia burgdorferi using high-throughput screening. Drug Des Devel Ther. 2016 Apr 1;10:1307-22. doi: 10.2147/DDDT.S101486. eCollection 2016. PMID 27103785
- [Background] Guerzoni S, Pellesi L, Pini LA, Caputo F. Drug-drug interactions in the treatment for alcohol use disorders: A comprehensive review. Pharmacol Res. 2018 Jul;133:65-76. doi: 10.1016/j.phrs.2018.04.024. Epub 2018 Apr 30. PMID 29719204
- [Background] Liegner KB. Disulfiram (Tetraethylthiuram Disulfide) in the Treatment of Lyme Disease and Babesiosis: Report of Experience in Three Cases. Antibiotics (Basel). 2019 May 30;8(2):72. doi: 10.3390/antibiotics8020072. PMID 31151194
- [Derived] Kuvaldina M, Preston J, McClellan D, Pavlicova M, Brannagan TH, Fallon BA. A pilot study of disulfiram for individuals with persistent symptoms despite prior antibiotic treatment for Lyme disease. Front Med (Lausanne). 2025 Apr 2;12:1549324. doi: 10.3389/fmed.2025.1549324. eCollection 2025. PMID 40265182
- See also: NIH website review of disulfiram's risk of liver toxicity — https://www.ncbi.nlm.nih.gov/books/NBK548103/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were no pre-assignment procedures in the protocol.
Period: Overall Study
Arm/Group | 8 Week Disulfiram | 4 Week Disulfiram
Started (Started means that participants signed consent and were randomized to study medication.) | 6 | 5
Start of the Medication | 5 | 4
Completed All 8 Weeks of Drug Treatment | 1 | 2
Completed All 10 Weeks of Assessments | 4 | 2
Completed | 4 | 2
Not Completed | 2 | 3
Not completed — Physician Decision | 1 | 1
Not completed — COVID related pause | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 8 Week Disulfiram | 4 Week Disulfiram | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.83 (13.78) | 37.8 (14.16) | 40 (13.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Fatigue Severity Scale (FSS)
Description: This is a psychometrically validated self-report measure of fatigue. This measure consists of 11 items inquiring about the severity of fatigue in different situations during the past week. Scores for each item range from 1 to 7, where 1 indicates strong disagreement and 7 strong agreement. Higher scores indicate higher levels of fatigue. A responder on the FSS is an individual whose FSS total score has decreased by 0.7 its when compared baseline to week 10 (or last observation carried forward); 0.7 refers to the minimally clinical significant difference (MCID) in change over time. We report the number of participants who reached a meaningful reduction in fatigue (equal or more than MCID).
Time Frame: Change will be assessed over a 10 week interval
Population: We conduct an intent to treat analysis which covers all enrolled and randomized patients who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 8 Week Disulfiram | 4 Week Disulfiram
Number analyzed (Participants) | 5 | 4
Participants | 4 | 2
Statistical Analysis 1: Comparison: 8 Week Disulfiram vs 4 Week Disulfiram; Test type: Superiority; Odds Ratio (OR) = 4, 95% CI 2-sided [.21 to 75.66]

2. Primary Outcome: Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF)
Description: The Q-LES-Q - SF is a self-reported questionnaire, with 16 items evaluating overall enjoyment and satisfaction with physical health, mood, work, household and leisure activities, social and family relationships, daily functioning, sexual life, economic status, overall well-being and medications. Responses are scored on a 5-point scale, where higher scores indicate better enjoyment and satisfaction with life (possible range 14-70). Fourteen summated items create the total Q-LES-Q - SF score. Two last items, about medications and overall life satisfaction, are considered independently. Meaningful improvement on the Q-LES-Q to is a change score between baseline and week 10 (or last observation carried forward) of at least 6.8 points; 6.8 refers to the minimally clinical significant difference (MCID) where a score equal to or greater than 6.8 points represents an improved quality of file. We report # with meaningful improvement.
Time Frame: Change will be assessed over a 10 week interval
Population: We conduct an intent to treat analysis which covers all enrolled and randomized patients who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 8 Week Disulfiram | 4 Week Disulfiram
Number analyzed (Participants) | 5 | 4
Participants | 2 | 2
Statistical Analysis 1: Comparison: 8 Week Disulfiram vs 4 Week Disulfiram; Test type: Superiority; Odds Ratio (OR) = .67, 95% CI 2-sided [0.05 to 9.47]

3. Secondary Outcome: The Short Form (36) Health Survey (SF-36) Physical Component Summary (PCS)
Description: The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. The 8 scales are-vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning mental health. Each scale is directly transformed into a 0-100 scale, the lower the score the more disability and the higher the score the less disability. We calculate the Physical Component Summary (PCS) (representing physical functioning) which represent the items in the SF-36 representing physical functioning (Ware, 2000); as in the sub scales, lower scores indicate greater disability.The norm-based estimate has a mean of 50 and a standard deviation of 10. We report the magnitude of the score change from baseline to week 10 (or the last observation carried forward (LOCF); negative change scores indicate improvement.
Time Frame: Change will be assessed over a 10 week interval
Population: We conduct an intent to treat analysis which covers all enrolled patients who received study drug.
Measure: Mean (Standard Deviation); unit: Score on scale (baseline minus LOCF)
Arm/Group | 8 Week Disulfiram | 4 Week Disulfiram
Number analyzed (Participants) | 5 | 4
Score on scale (baseline minus LOCF) | -5.183 (4.126) | -6.466 (5.374)

4. Secondary Outcome: General Symptom Questionnaire (GSQ-30)- Assess Multisystemic Symptom Burden
Description: This is a psychometrically validated 30 item self-report measure of symptom burden. The measure asks participants to rate how bothered they have been with a particular symptom over a 2-week time frame. Responses are made on 5-point Likert scale ranging from "not at all" to "very much" (scored 0-4); and the total score ranges from 0-120. Higher scores indicate more symptom severity. We report the magnitude of the score change (week 10 or last observation carried forward (LOCF)) minus the baseline score; a positive change score indicates improvement.
Time Frame: Change will be assessed over a 10 week interval
Population: We conduct an intent to treat analysis which covers all enrolled and randomized patients who received study drug.
Measure: Mean (Standard Deviation); unit: change in score (baseline minus LOCF)
Arm/Group | 8 Week Disulfiram | 4 Week Disulfiram
Number analyzed (Participants) | 5 | 4
change in score (baseline minus LOCF) | 25.6 (12.402) | 6.25 (20.790)

5. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS-29) Symptom Summary Score on Sleep Disturbance, Pain, Anxiety, Depression, and Low Energy/Fatigue (SPADE)
Description: The PROMIS-29 is a psychometrically validated 29 item self-report measure covering 7 domains. The questions are ranked on a 5-point Likert Scale. The composite score on 5 symptoms of the 7 domains is known as the SPADE summary score (sleep disturbance, pain, anxiety, depression, and low energy/fatigue); this represents the most common chronic symptoms in the general population. Each domain has 5 response options (e.g., 1=not at all to 5=very much), with scale scores ranging from 4 to 20 and higher scores indicating worse symptom severity. Using the scores from these 5 domains, we calculated the average score (SPADE score); the SPADE score ranges from 1 to 5 with higher scores indicating more symptom severity. We report the magnitude of the change in SPADE scores from baseline to week 10 (or the last observation carried forward (LOCF)); a positive change score indicates improvement.
Time Frame: Change will be assessed over a 10 week interval
Population: We conduct an intent to treat analysis which covers all enrolled and randomized patients who received study drug.
Measure: Mean (Standard Deviation); unit: Score on scale (baseline minus LOCF)
Arm/Group | 8 Week Disulfiram | 4 Week Disulfiram
Number analyzed (Participants) | 5 | 4
Score on scale (baseline minus LOCF) | 6.86 (3.71) | 5.95 (5.15)

6. Secondary Outcome: The Short Form (36) Health Survey (SF-36) Mental Component Summary (MCS)
Description: The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. The 8 scales are-vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning mental health. Each scale is directly transformed into a 0-100 scale, the lower the score the more disability and the higher the score the less disability. We calculate the Mental Component Summary (MCS) (representing physical functioning) which represent the items in the SF-36 representing physical functioning (Ware, 2000); as in the sub scales, lower scores indicate greater disability.. The norm-based estimate mean is 50 with a standard deviation of 10. We report the magnitude of the change in scores from baseline to week 10 (or the last observation carried forward (LOCF)); a negative change score indicates improvement.
Time Frame: Change will be assessed over a 10 week interval
Population: We conduct an intent to treat analysis which covers all enrolled and randomized patients who received study drug.
Measure: Mean (Standard Deviation); unit: Score on scale (baseline minus LOCF)
Arm/Group | 8 Week Disulfiram | 4 Week Disulfiram
Number analyzed (Participants) | 5 | 4
Score on scale (baseline minus LOCF) | -3.76 (15.437) | -4.814 (5.486)

ADVERSE EVENTS:
Time Frame: up to 14 weeks
Description: 11 patients signed consent and were randomized. 1 of these did not take any medication due to the onset of the COVID pandemic. 1 had data removed due to a later identified ineligibility.
Groups:
- 8 Week Disulfiram: Patients in this group receive disulfiram for 8 weeks. The dosing schedule is fixed-flexible, starting at 250 mg every other day at week 1, 250 mg daily for week 2, 250 mg alternating with 500 mg for week 3, and 500 mg daily for week 4 to week 8. Dose increases are based on clinical judgment guided by patient tolerance, response, body weight, and side effects.
  Disulfiram: Patients will receive disulfiram for 8 weeks .
- 4 Week Disulfiram: Patients in this group receive disulfiram for 4 weeks followed by placebo capsules for 4 weeks. The dosing schedule is fixed-flexible, starting at 250 mg every other day at week 1, 250 mg daily for week 2, 250 mg alternating with 500 mg during week 3, and 500 mg daily during week 4. Placebo capsules are given during weeks 5-8. Dose increases are based on clinical judgment guided by patient tolerance, response, body weight, and side effects.
  Disulfiram: Patients will receive disulfiram for 4 weeks followed by placebo for 4 weeks .
Arm/Group | 8 Week Disulfiram | 4 Week Disulfiram
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/5 | 1/4
Other Adverse Events (participants affected / at risk) | 5/5 | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 8 Week Disulfiram (N=5) | 4 Week Disulfiram (N=4)
ER visit (Immune system disorders) | 0 (0) | 1 (1) — 10 days after ending disulfiram treatment early (due to headaches), an episode of throat tightness nausea and light-headedness occurred. The patient (hx of asthma) went to ER and was treated for emerging possible anaphylaxis and recovered.
Short-term hospitalization (Hepatobiliary disorders) | 1 (1) | 0 (0) — Symptoms (severe abdominal pain) associated with elevated liver function tests led to a short-term hospitalization for evaluation. Episode probably related to a disulfiram reaction, but triggering exposure unclear; patient recovered.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 8 Week Disulfiram (N=5) | 4 Week Disulfiram (N=4)
Mild-moderately elevated liver function tests (Hepatobiliary disorders) | 3 (3) | 0 (0)
Mildly elevated serum creatinine (Renal and urinary disorders) | 1 (1) | 0 (0)
Moderate headache (General disorders) | 1 (1) | 0 (0)
Moderate to severe sore throat/throat hoarseness (General disorders) | 2 (2) | 0 (0)
Moderate to severe hypersomnia/sleepiness (General disorders) | 2 (2) | 0 (0)
Moderate tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Moderate shooting pain (Nervous system disorders) | 0 (0) | 1 (1)
Moderate neuromotor weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Moderate photosensitivity (Eye disorders) | 1 (1) | 0 (0)
Moderate dizziness (General disorders) | 1 (1) | 0 (0)
Moderate temperature fluctuations (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study did not reach its goal of 24 participants largely due to the impact of the COVID-19 pandemic on the ability to recruit subjects. Our small sample limits the conclusions that can be drawn from this trial, but the findings will be helpful to inform future studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-25): https://cdn.clinicaltrials.gov/large-docs/67/NCT03891667/Prot_SAP_000.pdf